CLINICAL TRIAL: NCT01441258
Title: Adaptation of Dialectical Behavior Therapy Skills-Groups for Individuals With Suicidal Ideation and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maurizio Fava, MD (Other)
Responsible Party: Sponsor-Investigator, Maurizio Fava, MD, Executive Vice Chair, Department of Psychiatry, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001088
Record Dates: First submitted 2011-09-21; First posted 2011-09-27 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Suicidal Ideation; Major Depressive Disorder
MeSH Terms: conditions — Suicidal Ideation; Depressive Disorder, Major | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical Behavior Therapy Skills (DBT-S) Groups (Experimental): Patients in the Dialectical Behavior Therapy Skills (DBT-S) group will receive the newly adapted 18-week group-skills training protocol, one-and-a-half hours in length, with weekly homework assignments to facilitate skill generalization.
  Interventions: Behavioral: Dialectical Behavior Therapy Skills (DBT-S) Groups
- Wait List-Treatment as Usual (Placebo Comparator): Participants assigned to the wait-list condition will be given the opportunity to participate in a DBT skills group after their 18-week wait period has ended.
  Interventions: Behavioral: Wait List-Treatment as Usual; Behavioral: No intervention-treatment as usual

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy Skills (DBT-S) Groups — The intervention will be delivered within an 18-week, once-weekly, one-and-half-hour skill group (8 participants per group) comprised of the same four modules administered in standard DBT skills training groups: (1) mindfulness, (2) interpersonal effectiveness, (3) emotion regulation, and (4) distress tolerance. There will be four sessions for each module totaling 16 sessions. There will be two booster sessions reviewing mindfulness and the concept of dialectics in-between each of the modules (i.e., between modules 2 and 3 and 3 and 4).
  Arms: Dialectical Behavior Therapy Skills (DBT-S) Groups
Behavioral: Wait List-Treatment as Usual — Participants will be seen by their standard treaters for 18 weeks as usual.
  Arms: Wait List-Treatment as Usual
Behavioral: No intervention-treatment as usual — Participants will receive the intervention after 18 weeks in the treatment as usual group.
  Arms: Wait List-Treatment as Usual

SUMMARY:
Harley and colleagues demonstrated that adding Dialectical Behavior Therapy (DBT) skills-groups and therapist consultation to treatment as usual successfully reduced symptoms of depression. The present study will expand upon these findings. Second, DBT is not known for reducing suicidal ideation (SI), a major risk factor for suicide . The present study will tailor the aforementioned skills-groups to specifically target suicidal thoughts and behaviors through Cognitive Behavior Therapy (CBT) strategies aimed at increasing problem-solving deficits, hopelessness, and negativistic thinking. Third, the present study will extend this DBT-based approach to a novel population. Fourth, the present study is the first DBT intervention to employ state-of-the-art multi-method measurement (including objective assessment) of suicidal thoughts and behaviors.

The investigators hypothesize that participants in the DBT skills (DBT-S) group will show improvements in level of suicidality as measured by decreased scores on the Beck Scale for Suicide Ideation as compared with participants in the Wait List-Treatment as Usual (WL-TAU) group.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be at least 18 years of age.
2. Participants will meet criteria for Major Depressive Disorder (MDD) on the Structured Clinical Interviews for Axis I DSM-IV Disorders
3. Participants must report current suicidal ideation on the Self-Injurious Thoughts and Behaviors Interview
4. Participants must have an outpatient psychiatric provider who they see "regularly" (i.e., at least every other week for therapy, case management, or medication management).
5. English language proficiency.

Exclusion Criteria:

1. DSM-IV diagnosis of bipolar disorder, schizophrenia, psychotic disorder NOS, or personality disorders.
2. Active current substance dependence.
3. Severe or unstable medical conditions that would prohibit regular group attendance or participation.
4. Other group therapy.
5. Significant dementia or cognitive impairment that would interfere with the learning of DBT skills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Beck Scale for Suicidal Ideation (SSI) | Participants will be assessed using the SSI monthly throughout the duration of their study participation for up to 15 months (see description for details)
  If randomized to the intervention, they will be assessed monthly for 18 weeks, then at 3 and 6-month follow-up visits. If they are randomized to the Wait list-Treatment as Usual (WL-TAU) group and then cross over into the intervention group, they will be assessed for a total of 36 weeks, not including the 3 and 6-month follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Maren Nyer, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Harley R, Sprich S, Safren S, Jacobo M, Fava M. Adaptation of dialectical behavior therapy skills training group for treatment-resistant depression. J Nerv Ment Dis. 2008 Feb;196(2):136-43. doi: 10.1097/NMD.0b013e318162aa3f. PMID 18277222
- [Background] Nock MK, Park JM, Finn CT, Deliberto TL, Dour HJ, Banaji MR. Measuring the suicidal mind: implicit cognition predicts suicidal behavior. Psychol Sci. 2010 Apr;21(4):511-7. doi: 10.1177/0956797610364762. Epub 2010 Mar 9. PMID 20424092